CLINICAL TRIAL: NCT05837013
Title: Comparison of Open and Laparoscopic Total Extraperitoneal Inguinal Hernia Repair (TEP) Performed Under Blocked Spinal Anesthesia and General Anesthesia: Prospective Randomized Study
Brief Title: Open and Laparoscopic Total Extraperitoneal Repair Under Spinal Anesthesia Versus General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Collaborators: Van Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Eşref Ulutaş, Principal Investigator, Konya City Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 33333333
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Pain, Postoperative; Postoperative Complications; Inguinal Hernia
Keywords: spinal anesthesia; inguinal Hernia; general anesthesia; laparoscopic total extraperitoneal repair
MeSH Terms: conditions — Pain, Postoperative; Postoperative Complications; Hernia, Inguinal | interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- General anesthesia (GA) and TEP Group (Experimental): General anesthesia: No premedication will be applied. In the waiting room, 10 mL/kg of Ringer's lactate solution will be infused IV in 30 minutes. In Group I, 2-2.5 mg/kg propofol and 1 μg/kg fentanyl IV will be given for induction; 0.6 mg/kg rocuronium will then be used to provide the muscle relaxation needed for intubation. After intubation, the tidal volume will be set to 6-8 mL/kg and the respiratory frequency PetCO2 32-36 mmHg in volume-controlled ventilation (VCV) mode. Anesthesia will continue to be provided with sevoflurane (1.5%-2%), oxygen-air mixture (FiO 2 = 0.4) and repeated doses of rocuronium (0.015 mg/kg). At the end of the surgery, neostigmine (2-2.5 mg) and atropine (1 mg) will be given IV to antagonize the residual neuromuscular block.
  Interventions: Procedure: General anesthesia (GA)
- Spinal anesthesia (with nerve block) (SA) and TEP Group (Active Comparator): Spinal Anesthesia and Nerve Block: No premedication will be applied. Spinal anesthesia will be administered to the patients in this group in the sitting position with a 27G Quincke needle (15 mg hyperbaric 0.5% bupivacaine) to be entered through the L2-L3 or L3-L4 interval. If hypotension develops, it will be corrected with a crystalloid infusion and ephedrine. These patients will be administered intravenous sedation with increasing doses of midazolam to provide adequate sedation. According to Hadzic, II and IH nerve block will be performed by applying 10 mL of 0.75% ropivacaine 2 cm above and 2 cm medial to the anterior superior iliac spine.
  Interventions: Procedure: Spinal anesthesia (with nerve block)
- General anesthesia (GA) and open surgical procedure (Lichtenstein) (Experimental): General anesthesia: No premedication will be applied. In the waiting room, 10 mL/kg of Ringer's lactate solution will be infused IV in 30 minutes. In Group I, 2-2.5 mg/kg propofol and 1 μg/kg fentanyl IV will be given for induction; 0.6 mg/kg rocuronium will then be used to provide the muscle relaxation needed for intubation. After intubation, the tidal volume will be set to 6-8 mL/kg and the respiratory frequency PetCO2 32-36 mmHg in volume-controlled ventilation (VCV) mode. Anesthesia will continue to be provided with sevoflurane (1.5%-2%), oxygen-air mixture (FiO 2 = 0.4) and repeated doses of rocuronium (0.015 mg/kg). At the end of the surgery, neostigmine (2-2.5 mg) and atropine (1 mg) will be given IV to antagonize the residual neuromuscular block.
  Interventions: Procedure: General anesthesia (GA)
- Spinal anesthesia (with nerve block) (SA) open surgical procedure (Lichtenstein) (Active Comparator): Spinal Anesthesia and Nerve Block: No premedication will be applied. Spinal anesthesia will be administered to the patients in this group in the sitting position with a 27G Quincke needle (15 mg hyperbaric 0.5% bupivacaine) to be entered through the L2-L3 or L3-L4 interval. If hypotension develops, it will be corrected with a crystalloid infusion and ephedrine. These patients will be administered intravenous sedation with increasing doses of midazolam to provide adequate sedation. According to Hadzic, II and IH nerve block will be performed by applying 10 mL of 0.75% ropivacaine 2 cm above and 2 cm medial to the anterior superior iliac spine.
  Interventions: Procedure: Spinal anesthesia (with nerve block)

INTERVENTIONS:
Procedure: Spinal anesthesia (with nerve block) — Spinal Anesthesia and Nerve Block: No premedication will be applied. Spinal anesthesia will be administered to the patients in this group in the sitting position with a 27G Quincke needle (15 mg hyperbaric 0.5% bupivacaine) to be entered through the L2-L3 or L3-L4 interval. If hypotension develops, it will be corrected with a crystalloid infusion and ephedrine. These patients will be administered intravenous sedation with increasing doses of midazolam to provide adequate sedation. According to Hadzic, II and IH nerve block will be performed by applying 10 mL of 0.75% ropivacaine 2 cm above and 2 cm medial to the anterior superior iliac spine.
  Arms: Spinal anesthesia (with nerve block) (SA) and TEP Group; Spinal anesthesia (with nerve block) (SA) open surgical procedure (Lichtenstein)
Procedure: General anesthesia (GA) — General anesthesia: No premedication will be applied. In the waiting room, 10 mL/kg of Ringer's lactate solution will be infused IV in 30 minutes. In Group I, 2-2.5 mg/kg propofol and 1 μg/kg fentanyl IV will be given for induction; 0.6 mg/kg rocuronium will then be used to provide the muscle relaxation needed for intubation. After intubation, the tidal volume will be set to 6-8 mL/kg and the respiratory frequency PetCO2 32-36 mmHg in volume-controlled ventilation (VCV) mode. Anesthesia will continue to be provided with sevoflurane (1.5%-2%), oxygen-air mixture (FiO 2 = 0.4) and repeated doses of rocuronium (0.015 mg/kg). At the end of the surgery, neostigmine (2-2.5 mg) and atropine (1 mg) will be given IV to antagonize the residual neuromuscular block.
  Arms: General anesthesia (GA) and TEP Group; General anesthesia (GA) and open surgical procedure (Lichtenstein)

SUMMARY:
Inguinal hernia surgery is one of the most frequently performed procedures among general surgery cases. As with many open surgical methods, this repair is also performed laparoscopically. Among these closed methods, the most frequently applied method is laparoscopic total extraperitoneal repair (TEP). In general, this surgery is performed under general anesthesia (GA) in many centers. However, in cases where general anesthesia is inconvenient, local or other anesthesia methods are preferred.

It has been stated in many studies in the literature that this surgery can be performed with methods other than general anesthesia. In a study of 480 patients, one of which was Sinha et al., it was shown that this surgical procedure was successfully performed under spinal anesthesia (SA).

In a prospective randomized study by Dönmez et al., patients who underwent TEP under general anesthesia and spinal anesthesia were compared. It has been reported that TEP repair can be performed safely under SA and that SA is associated with less postoperative pain, better recovery, and better patient satisfaction than GA.2 In a retrospective study by Yıldırım et al. It has been shown that there is significantly less need for analgesics and better patient satisfaction.

There are also many meta-analyses made on this subject in the literature. Compared with GA in these, SA was associated with a longer operative time, and postoperative pain and nausea and vomiting were less in SA. However, the risk of urinary retention in SA was significantly increased. It was observed that there was no significant difference in surgical complications such as seroma and wound infection.

Despite all these studies, until now, there is no clear consensus on which anesthesia should be used.

The aim of the study is to show the effect of both the surgical method and the anesthesia method on the patient during surgery and in the early postoperative period in inguinal hernia

DETAILED DESCRIPTION:
Patients who underwent laparoscopic total extraperitoneal (TEP) inguinal hernia repair and open surgical procedure (Lichtenstein) with the diagnosis of inguinal hernia will be divided into 2 groups. General anesthesia (GA) will be applied to the 1st group, and ileoinguinal (II) and ileohypogastric (IH) nerve block together with spinal anesthesia (SA) to the 2nd group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with inguinal hernias.
* Over 18 years old

Exclusion Criteria:

* Younger than 18 years
* Those who have had previous abdominal surgery,
* Incarcerated or strangulated inguinal hernias,
* Recurrent hernias,
* Coagulopathies,
* Patients with musculoskeletal deformity,
* Those with chronic pain,
* Those who use drugs that affect the central nervous system daily,
* Those with a body mass index (BMI) over 40 kg/m2,
* Patients with contraindications to the recommended anesthetic technique.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | Postoperative 24 hours
  It will be measured using the Visual Analog Score (VAS). The patient will be asked to choose between the number 1 with the least pain and the number 10 with the most pain. The lowest score on this scale is 1, and the highest score is 10.

SECONDARY OUTCOMES:
Adverse postoperative events | Postoperative 24 hours
  headache, nausea/vomiting, anxiety, abdominal discomfort and urinary retention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Science Van Training and Research Hospital, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sinha R, Gurwara AK, Gupta SC. Laparoscopic total extraperitoneal inguinal hernia repair under spinal anesthesia: a study of 480 patients. J Laparoendosc Adv Surg Tech A. 2008 Oct;18(5):673-7. doi: 10.1089/lap.2007.0219. PMID 18803509
- [Background] Donmez T, Erdem VM, Sunamak O, Erdem DA, Avaroglu HI. Laparoscopic total extraperitoneal repair under spinal anesthesia versus general anesthesia: a randomized prospective study. Ther Clin Risk Manag. 2016 Oct 27;12:1599-1608. doi: 10.2147/TCRM.S117891. eCollection 2016. PMID 27822053
- [Background] Yildirim D, Hut A, Uzman S, Kocakusak A, Demiryas S, Cakir M, Tatar C. Spinal anesthesia is safe in laparoscopic total extraperitoneal inguinal hernia repair. A retrospective clinical trial. Wideochir Inne Tech Maloinwazyjne. 2017 Dec;12(4):417-427. doi: 10.5114/wiitm.2017.72325. Epub 2017 Dec 29. PMID 29362658
- [Background] Li L, Pang Y, Wang Y, Li Q, Meng X. Comparison of spinal anesthesia and general anesthesia in inguinal hernia repair in adult: a systematic review and meta-analysis. BMC Anesthesiol. 2020 Mar 10;20(1):64. doi: 10.1186/s12871-020-00980-5. PMID 32156258
- [Background] Hajibandeh S, Hajibandeh S, Mobarak S, Bhattacharya P, Mobarak D, Satyadas T. Meta-Analysis of Spinal Anesthesia Versus General Anesthesia During Laparoscopic Total Extraperitoneal Repair of Inguinal Hernia. Surg Laparosc Endosc Percutan Tech. 2020 Aug;30(4):371-380. doi: 10.1097/SLE.0000000000000783. PMID 32217883